CLINICAL TRIAL: NCT06518148
Title: Causes of Visual Impairment Among Patients Applying for the Visually Disability Certification in Upper Egypt: A Retrospective Study
Brief Title: Causes of Visual Impairment Among Patients Applying for the Visually Disability Certification
Status: Active, not recruiting | Type: Observational
Sponsor: New Valley University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Kamel Ahmed Hassan, Lecture of ophthalmology ,faculty of medicine , new valley university, New Valley University
Other Study IDs: CVIAPAVDCUE
Record Dates: First submitted 2024-07-14; First posted 2024-07-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders | interventions — Evoked Potentials, Visual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 1- uncorrected and best corrected visual acuity (UCVA and BCVA) by Snellen's-chart.2-slit lamp bio microscopy (Haag-Streit, USA).3-IOP measurements (Goldmann Applanation tonometer) — diagnostic test;UCVA, IOP, Electrophysiological study
  Other Names: 3-fundus examination (+90D lens and indirect ophthalmoscope).; 4- Electrophysiological study visual evoked potential (VEP) and full filed electroretinogram (Metrovision machine).

SUMMARY:
Causes of Visual Impairment Among Patients Applying for the Visually Disability Certification in Upper Egypt: A Retrospective Study

DETAILED DESCRIPTION:
There are at least 2.2 billion individuals with near- or far-sightedness worldwide. Nearly half of these cases-at At least 1 billion-have untreated vision impairment that may have been avoided. The leading cause of blindness or impaired distant vision among these 1 billion people is diabetic retinopathy (3.9 million), age-related macular degeneration (8 million), cataracts (94 million), refractive error (88.4 million), and glaucoma (7.7 million). Presbyopia (826 million) is the primary ailment that impairs close vision.

According to estimates, there are four times as many cases of distant vision impairment in low- and middle-income areas as there are in high-income areas.

Aging populations and population expansion are predicted to raise the likelihood that more people may have visual impairment. Early on, irreversible severe visual impairment in young children can lead to delayed motor, verbal, emotional, social, and cognitive development, which can have long-term effects. Children of school age who are visually impaired may also perform less academically. The quality of life is significantly impacted by vision impairment in adult populations. Adults who are visually impaired may have greater rates of anxiety and depression as well as decreased employment rates.

Vision impairment in older persons can increase their risk of falling and breaking bones, walking difficulties, social isolation, and early admission into nursing homes or other care facilities.

According to estimates, vision impairment costs the world's economy $411 billion annually in lost productivity (purchasing power parity) . This amount is greatly above the predicted $25 billion cost gap incurred from treating vision impairment.

This study is to demonstrate the causes of visual impairment in upper Egypt among the different age groups and evaluate the possibility of preventing these disorders

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to The Ministry of Social Solidarity with visual Disability in upper Egypt who were examined in the visual disability screening program from 2020-2024.

Exclusion Criteria:

* The patients who had decreased vision but did not fit with the WHO definition of visual disability.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to The Ministry of Social Solidarity with visual Disability in upper Egypt who were examined in the visual disability screening program from 2020-2024-no age or gender limits for the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The relative frequencies or prevalence of different eye diseases/conditions causing visual disability | 10 month
2-Ranking of the leading cause(s) of visual impairment | 10 month

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
we share in a multicenter study.